CLINICAL TRIAL: NCT02109055
Title: Application of Exercises Based on the Pilates Method on the Functional Capacity in Postoperative Surgery Coronery Artery Bypass Grafting: Randomized Clinical Trial
Brief Title: Application of Exercises Based on the Pilates in Coronary Artery Bypass Grafting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Rodrigo Della Méa Plentz, PhD, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PILATESCRM1
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular Diseases; Thoracic Surgery; Exercise Therapy
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pilates (Experimental): Regarding upper limb exercises the limit of flexion and abduction less than 90°, with the exercises involving only the movement of flexion and extension of elbow shoulder will be respected. Along with patient data will be an exercise protocol based on the Pilates method that will be performed by a trained team of physiotherapists. Before and after the exercises the data of heart rate, blood pressure, oxygen saturation and subjective feeling of perceived exertion using the Modified Borg scale will be listed.
  Interventions: Other: Pilates
- Convencional Physiotherapy (Active Comparator): The conventional physiotherapy group will continue with the routine hospital consisting of respiratory physiotherapy.
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Pilates — The exercise program will be held during the period of hospitalization for six days, often two to three sessions per day, totaling 12 sessions.
  Arms: Pilates
Other: Conventional Physiotherapy — The conventional physiotherapy group will continue with the routine hospital consisting of respiratory physiotherapy, twice daily, six days.
  Arms: Convencional Physiotherapy

SUMMARY:
The major cause of mortality worldwide is due to cardiovascular diseases. A way to treat these diseases is coronary artery bypass grafting, one of the most common surgical procedures in the world. The incidence of post-operative complications contributes to functional decline of the patient, reduced quality of life and post-discharge mortality. Also, cardiac surgery leads to changes in lung capacity and respiratory muscle strength, causing a decrease in the function lung. Physical therapy proves to be an effective tool to combat changes resulting from cardiac surgery, demonstrating beneficial results in the pulmonary function, functional capacity, and peripheral and respiratory muscle strength. The Pilates method has been studied as a therapeutic way to healthy subjects and various kinds of diseases, but there are no studies in the literature evaluating the effect method in patients after coronary artery bypass surgery.

The aim of this study is to investigate the effect of Pilates on functional capacity , flows and lung volumes, respiratory and peripheral muscle strength after coronary artery bypass grafting.

Randomized clinical trial in which patients will be eligible after elective coronary artery bypass surgery, randomly allocated into two groups : conventional physiotherapy group (n = 15) and Pilates method associated with conventional physiotherapy group (n = 15). The outcomes will be assessed by blinded evaluator and data randomization will be performed through by electronic randomization.The interventions will take place during the length of stay in the hospital, totalizing a maximum of six days of intervention.

It is expected that the application of the Pilates method exercise method associated with conventional physiotherapy in patients in postoperative coronary artery bypass grafting improves functional capacity, flows and lung volumes and respiratory and peripheral muscle strength.

DETAILED DESCRIPTION:
The exercise program will be held during the period of hospitalization for six days, often two to three sessions per day, totaling 12 sessions. The intervention will start on the first day postoperatively. The program may not exceed 30% of maximum heart rate reserve of the patient that will be calculated by the Karvonen formula (Karvonen, Kentala et al., 1957). The exercises will be conducted at the patient's bedside, using light resistance springs representing the lowest possible burden of springs to be used in the Pilates method. The exercises will be performed on the upper limbs alternating between the left and right upper limb and likewise would run with the lower limbs by means of a protocol consists of four exercises until the limit of resistance of the patient or interrupt pre-established criteria.

One set of each exercise with a range of up to two minutes between exercises will be held. In the first three days of intervention 10 repetitions of each exercise and the remaining three days a total of 15 repetitions of each movement will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Individuals in postoperative coronary artery bypass grafting, extubated within 24 hours after surgery, hemodynamically stable, with no ischemic changes and/or complex arrhythmias on electrocardiogram e who have performed the first surgery and surgery alone.

Exclusion Criteria:

* Patients with decompensated heart failure, presence of any comorbidity, such as unstable angina, associated neurological disease, moderate to severe respiratory illness prior diagnosed by the attending physician, acute respiratory dysfunction in the post - operative, active infectious disease or fever; vascular disease disabling peripheral, unstable ventricular arrhythmia; musculoskeletal disease that limits the practice of Pilates will be excluded.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-12 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of functional capacity | six days

SECONDARY OUTCOMES:
Evaluation of respiratory muscle strength | six days
Evaluation of respiratory volumes and flows | six days
Evaluation of peripheral muscle strength | six days

CONTACTS AND LOCATIONS:
Overall Officials: Manoela H dos Reis, Graduated, Study Chair — Federal University of Health Science of Porto Alegre; Leonardo F Neves, Graduated, Study Chair — University of the Sinos Valley; Cinara Stein, Master, Study Chair — Federal University of Health Science of Porto Alegre; Mirelle Hugo, Undergrad, Study Chair — Federal University of Health Science of Porto Alegre; Aline Miozzo, Graduated, Study Chair — Universidade Federal de Santa Maria; Christian Coronel, Master, Study Chair — Instituto de Cardiologia do Rio Grande do Sul
Locations (1):
- Rodrigo Della Méa Plentz, Porto Alegre, Rio Grande do Sul, Brazil